CLINICAL TRIAL: NCT04281693
Title: Identification of a New Screening Strategy for 2019 Novel Coronavirus Infection
Brief Title: A New Screening Strategy for 2019 Novel Coronavirus Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 307-nCoV
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Novel Coronavirus Infection Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening participants (Experimental)
  Interventions: Diagnostic Test: Standard screening strategy; Diagnostic Test: New screening strategy

INTERVENTIONS:
Diagnostic Test: Standard screening strategy — The pharyngeal swab specimen was obtained and sent for NCIP RNA detection by individual testing.
Diagnostic Test: New screening strategy — The pharyngeal swab specimen was obtained and sent for NCIP RNA detection by minipool testing.

SUMMARY:
Since Dec 2019, over 70000 novel coronavirus infection pneumonia (NCIP) patients were confirmed. 2019 novel coronavirus (2019 nCoV) is a RNA virus, which spread mainly from person-to-person contact. Most of the symptoms are non-specific, including fever, fatigue, dry cough. Sever NCIP patients may have shortness of breath and dyspnea, and progress to acute respiratory distress syndrome (ARDS) and multiple organ dysfunction syndrome (MODS). The mortality is reported to be around 2.3%. Thus, early detection and early treatment is very important to the improvement of NCIP patients' prognosis. At present, NCIP RNA detection of pharyngeal swab specimen by RT-PCR is recommended. However, due to the universal susceptibility to 2019 nCoV in general population and limited number of NCIP RNA detection kits available, to identify an efficient screening strategy is urgently needed. This study aim to develop and validate the diagnostic accuracy and screening efficiency of a new NCIP screening strategy, which can benefit the disease prevention and control.

DETAILED DESCRIPTION:
This clinical trial is designed to compare the screen accuracy and efficiency of two screening strategies. Considering that the general population is susceptible to 2019 nCoV, a great number of people need to be screened for NCIP. The new screening strategy of minipool testing may not only obtain a comparable accuracy to the standard individual testing, but also save time and money, which may benefit the current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Who agree to participate in the study and sign written informed consent

Exclusion Criteria:

* Confirmed NCIP patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Screening accuracy | 1 month
  The screening accuracy of the two screening strategies were calculated and compared.

SECONDARY OUTCOMES:
Cost-effectiveness analysis | 1 month
  The costs of the two screening strategies were recorded. Cost-effectiveness analysis were performed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Principal Investigator — Beijing 302 Hospital
Locations (1):
- the Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853